CLINICAL TRIAL: NCT00359580
Title: Genetic Studies in the Amish and Mennonites
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970192; 97-HG-0192
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-06-27

CONDITIONS: Genetic Disease
Keywords: Rare Diseases; Consanguinity; Natural History
MeSH Terms: conditions — Genetic Diseases, Inborn; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AGDB: Those individuals who are listed in the Fisher Family History and other genealogy books ordatabases will be included in the AGDB.

SUMMARY:
The purposes of this study are to identify the genes responsible for several inherited disorders commonly seen in the Amish and Mennonite populations and learn more about the natural history (medical problems that develop over time) of these disorders. In addition, researchers will establish a computer database containing Amish genealogies, derived largely from the community s extensive records of births, marriages, deaths, etc., that will help construct pedigrees (family trees) for genetic study.

The Amish and Mennonite peoples have a high rate of intermarriage within their individual communities, with a resulting high incidence of inherited disorders. Many of these disorders, such as cartilage-hair hypoplasia, Ellis-van Creveld syndrome, and others, are rarely seen outside these communities. New research using state-of-the-art methodologies in genetics will add to current knowledge about the causes and symptoms of these disorders that will eventually aid in their diagnosis and medical management.

Patients with inherited disorders that occur frequently in the Amish and Mennonite populations and their family members may be eligible for this study. Individuals from both within and outside these communities may enroll.

Participants will be evaluated with a review of their medical records and their personal and family medical history and a brief physical examination. A small tissue sample will be collected for genetic studies. This will be either a blood sample (3 teaspoons from adults and 1 to 3 teaspoons from children, depending on their size) or a mouth swab (cells removed from inside the cheek by gentle brushing). Some participants may undergo additional procedures, such as diagnostic X-rays, brain scans, echocardiogram (heart ultrasound) or other studies.

If genetic testing shows a gene change (mutation), the participant will be notified to that effect in writing and offered counseling in their home regarding the test results and their implications....

DETAILED DESCRIPTION:
The Amish and Mennonite populations represent outstanding communities for the study of genetic disease for a number of reasons. There is a high degree of inbreeding, resulting in a high frequency of recessive disorders, many of which are seen rarely or are unknown outside of this population. Extensive genealogical records are available, and the average family size is large. This proposal includes a number of collaborators who have had extremely close, extensive interaction with the Lancaster County Amish over the past decade; their relationships with the community are invaluable to the success of this project. We have had substantial success with this research over the past seven years, leading to the discovery of the molecular etiology of four human diseases and the establishment of a useful database and tools for genealogical analysis. We propose to continue this line of research to further characterize these disorders and identify additional ones, as well as enlarging a computerized Anabaptist genealogy.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects are divided into two groups:

Group A:

Patients and their families with known or suspected Mendelian or complex traits, who will be enrolled in the molecular genetics and phenotypic characterization study.

Informed consent will be obtained from each of these subjects.

Group B:

Those individuals who are listed in the Fisher Family History and multiple other genealogy books will be included in the AGD database.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2004-02-10 (Actual)

PRIMARY OUTCOMES:
Database | Ongoing
  To maintain, expand, and use an electronic database containing the Anabaptist genealogies to facilitate the generation of pedigrees and calculation of common ancestors between nuclear families.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie G Biesecker, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Clinic for Special Children, Strasburg, Pennsylvania

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1997-HG-0192.html